CLINICAL TRIAL: NCT05234229
Title: Influenza and Pertussis Vaccination Status of Women in Immediate Postpartum and Caregivers in the Maternity Hospital of Nancy
Brief Title: Influenza and Pertussis Vaccination Status of Women in Immediate Postpartum and Caregivers
Acronym: COVAGRIP
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: 2021PI087
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Pertussis/Whooping Cough; Influenza Viral Infections
Keywords: immunization; cocooning
MeSH Terms: conditions — Whooping Cough | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covagrip women in immediate post partum: women in immediate post partum
  Interventions: Other: Survey
- Caregivers: health care personnel
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Collection of immunization status by questionnaire

SUMMARY:
Pertussis is a bacterial respiratory infection caused by Bordetella pertussis. Highly contagious, it is potentially serious and even fatal in infants under 6 months of age. The immunity acquired through vaccination is very limited in time, requiring regular booster shots. There is a passive protection of the newborn by the maternal-fetal transmission of maternal antibodies, but it is brief. The infant's first vaccination is given at 2 months of age and immunity is not acquired until the second injection at 4 months of age. The booster at 11 months of age is essential to prolong this immunity.

In order to protect infants under 6 months of age, France has recommended since 2004 the cocooning strategy, which consists of vaccinating people likely to be in close contact with the infant during this period. This vaccination is therefore proposed to adults who are planning to have children, to the entourage of pregnant women, and in the immediate post-partum period for the mother (and people who were not vaccinated during pregnancy). This strategy was put in place following the international recommendation of a forum of scientific experts, the Global Pertussis Initiative.

In France, vaccination against pertussis is not currently recommended during pregnancy. There is no contraindication to vaccination during pregnancy and it is recommended in many countries.

Influenza is a viral respiratory infection caused by Myxovirus influenzae, which is highly contagious.

In France, vaccination against influenza is recommended for pregnant women, regardless of the trimester of pregnancy. It is also recommended for the entourage of infants under 6 months of age with risk factors for severe influenza.

There are few recent data in the scientific literature regarding influenza and pertussis vaccination coverage among pregnant or postpartum women in France. In addition, the COVID19 pandemic has recently reopened the debate on vaccination of the general population and caregivers. Knowing the current status of vaccination coverage among pregnant women and caregivers, their knowledge and fears regarding vaccination could help improve the information provided by healthcare staff.

ELIGIBILITY:
Inclusion Criteria:

* Person having received complete information about the research and not opposed to the study.
* Hospitalization in the post-partum service and within the last 5 days of delivery.
* women. caregivers

Exclusion Criteria:

* Female under 18 years of age,
* Woman under legal protection,
* Delivery of a stillborn child,
* Premature delivery < 35GA,
* Hospitalized newborn,
* Women who doesn't speak french.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18 years old, delivery after 35GA and healthcare staff of the University Maternity Hospital of Nancy in 2022. Person having received complete information about the research and not opposed to the study.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of influenza vaccination | 4 months
  To determine the rate of influenza immunization in immediate postpartum women and caregivers at the Nancy University Maternity Hospital in 2022 .
Prevalence of pertussis vaccination | 4 months
  To determine the rate of pertussis immunization in immediate postpartum and caregivers at the Nancy University Maternity Hospital in 2022

SECONDARY OUTCOMES:
awareness of own vaccination status | 4 months
  To determine the awareness of own vaccination status (yes; no; unknown) in immediate postpartum women regarding their influenza and pertussis immunization
Knowledge about vaccination | 4 months
  To determine the rate of right answers to a questionnaire about knowledge of influenza and pertussis vaccination, and the possibility of vaccination during pregnancy.
opinion on vaccination during pregnancy | 4 months
  To determine the rate of differences in vaccination coverage and knowledge among postpartum women and healthcare staff.
readiness to receive pertussis and influenzae immunization | 4 months
  to answer the readiness (yes; no; already vaccinated) to receive immunization after answering the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel HASCOET, Study Director — Maternité Régionale Universitaire CHRU NANCY
Locations (1):
- Maternite Regionale Universitaire CHRU NANCY, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No